CLINICAL TRIAL: NCT02995317
Title: The ≥65 Years NOrthern Jutland Cohort of Fall Risk Assessment With Objective Measurements (the NOCfao Study)
Brief Title: Who is Falling? - Fall Risk Prediction Among Community Dwelling Elderly.
Acronym: NOCfao
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College of Northern Denmark (Other)
Collaborators: Aalborg Municipality (Other); Aalborg University (Other)
Responsible Party: Sponsor
Other Study IDs: FOU-UU-006
Record Dates: First submitted 2016-12-13; First posted 2016-12-16 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Accidental Fall
Keywords: Aged; Gait; Postural Balance; Accelerometry; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Fall accidents
  Interventions: Other: Number of falls based on an one year follow-up

INTERVENTIONS:
Other: Number of falls based on an one year follow-up

SUMMARY:
The purpose of this study is to investigate if the level of physical activity, selected physical and psychological risk factors can predict risk of falling in older (≥65) community dwellers.

ELIGIBILITY:
Inclusion Criteria:

* Home dwelling
* Manage body transfer independently
* Walking ability for at least 10 meters with or without assistive devices

Exclusion Criteria:

* Progressive neurological or rheumatologically illness
* Diagnosed vestibular problems
* Experienced pain in a substantial degree, limiting or obstructing everyday living
* Known uncorrected visual or hearing problems.
* Serious difficulties in speaking, understanding or reading Danish.
* Cognitive impairment equivalent to Mini Mental State Examination < 23

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The study will be undertaken in Aalborg Municipality at different activity-centers and nursing homes in collaboration with care workers, nurses and staff at the activity centers, all employed at the Department of Elderly and Health. Furthermore the project manager arranges briefing meetings with groups of employees in order to provide clarification of the project and encourage support of the recruitment of the study-population. Participants satisfying the inclusion and exclusion criteria is contacted by the project group, to ensure that they fully understand what it takes to participate. Subsequently, an appointment for completion of the baseline data is made.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Self-reported number of falls confirmed by monthly phone calls | One year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bo Grarup, Principal Investigator — University College of Northern Denmark
Locations (1):
- University College of Northern Denmark, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Villumsen M, Grarup B, Christensen SWMP, Palsson TS, Hirata RP. "Study protocol for the >/=65 years NOrthern jutland Cohort of Fall risk Assessment with Objective measurements (the NOCfao study)". BMC Geriatr. 2020 Jun 8;20(1):198. doi: 10.1186/s12877-020-01535-6. PMID 32513121